CLINICAL TRIAL: NCT06377163
Title: Bacterial Pathogens Associated With Community-acquired Pneumonia in Children
Status: Completed | Type: Observational
Sponsor: Delta University for Science and Technology (Other)
Responsible Party: Principal Investigator, Amira Hussin Hussin Mohammed, Assistant professor at faculty of physical therapy, Delta University for Science and Technology
Other Study IDs: acquired pneumonia in children
Record Dates: First submitted 2024-04-10; First posted 2024-04-22 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Children Chest Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pediatric community acquired pneumonia (CAP) is one of the most common reasons for hospital admission, there is no reliable way of distinguishing the causative organism based on clinical features.

This study examined common pathogens of community-acquired pneumonia from 28 days up to 10 years in Dakahlia Governorate.

ELIGIBILITY:
- Inclusion criteria:

* Infants and children aged 28 days to ten years (male and female sexes).
* Patients diagnosed with community-acquired pneumonia.
* Pneumonia was diagnosed if the patient fulfilled has fever (temperature ≥38.3° C), Fast breathing (40 breaths per minute if the child is 1 year up to 10 years old), respiratory distress (tachypnea, retractions) and chest indrawing and cyanosis with compatible chest x-ray findings.

Exclusion criteria:

* Neonates
* Children more than 10 years
* Hospital acquired pneumonia
* Chronic lung disease, immunodeficiency and other congenital anomalies

Ages: 28 Days to 10 Years | Sex: All
Age Groups: Child
Study Population: A representative sample of 100 participants was taking by simple random sampling technique from children diagnosed to have community acquired pneumonia from Al Mansoura university hospital and Mansura International Hospital.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Complete blood count | At the baseline evaluation
  From each participant, a sample of 4 ml of fresh venous blood was collected from the peripheral vein by the sterile venipuncture technique & drawn into a vacuumed purple top tube containing an anticoagulant. It was performed using a fully automated hematology analyzer. This test measures the amounts and sizes of red blood cells, hemoglobin, white blood cells, and platelets. It will be aggregated to arrive at one report. Hemoglobin is usually reported in units of grams per liter, or grams per deciliter. The analyzer counts red blood cells, reporting the result in units of 106 cells per microliter of blood or 1012 cells per liter, and measures their average size, which is called the mean cell volume and expressed in femtoliters or cubic micrometers. The total white blood cell count is usually reported in cells per microliter of blood, or 109 cells per liter. The platelet count can be reported in units of cells per microliter of blood, 103 cells per microliter, or 109 cells per liter.
C-reactive protein (CRP) | At the baseline evaluation
  It was measured quantitatively in human serum by Beckman-Coulter AU Analyzers (USA).
  Sample preparation: 2 ml of blood in a sterile tube was centrifuged, then used immediately for CRP. C-reactive protein (CRP) is an annular (ring-shaped) pentameric protein found in blood plasma whose circulating concentrations rise in response to inflammation. Traditional CRP measurement only detected CRP in the range of 10 to 1,000 mg/L, whereas high-sensitivity CRP (hs-CRP) detects CRP in the range of 0.5 to 10 mg/L.
Blood culture and sensitivity on admission | At the baseline evaluation
  It was done using the BD Bactec 9050 Blood Culture System (USA, Catalog No. 445800) instrument. A culture was considered positive if any organism was identified.
Gastric lavage culture or sputum culture on admission | At the baseline evaluation
  It was inserted through the nose and down the stomach after nebulization with hypertonic saline at 5% for 10 seconds. Suction was applied for up to 15 seconds to collect the swallowed sputum in a sterile container. A culture was considered positive if any organism was identified.

CONTACTS AND LOCATIONS:
Locations (1):
- Amira Hussin Mohammed, Gamasa, Egypt

IPD SHARING:
Plan to Share IPD: Undecided